CLINICAL TRIAL: NCT01153243
Title: Does Administration of Vitamin D in African Americans With Hypovitaminosis D and Type 2 DM Improve Inflammatory Markers of Cardiovascular Disease?
Brief Title: Vitamin D and Inflammatory Markers of Cardiovascular Disease in African Americans With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cook County Health (Other Government)
Collaborators: Rush University (Other)
Responsible Party: Leon Fogelfeld MD, John H Stroger Hospital of Cook County
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #07-061
Record Dates: First submitted 2010-03-23; First posted 2010-06-30 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2009-03

CONDITIONS: Vitamin D Deficiency; Diabetes
Keywords: inflammatory markers
MeSH Terms: conditions — Vitamin D Deficiency; Diabetes Mellitus | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergocalciferol (Active Comparator): The investigators will give intervention group 12 weeks of Vitamin D (ergocalciferol 50,000 units every week)
  Interventions: Drug: Ergocalciferol
- Placebo pill (Placebo Comparator): The investigators will give intervention group 12 weeks of placebo pill (in pill every week)
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Ergocalciferol — Active Comparator: Ergocalciferol
  The investigators will give intervention group 12 weeks of Vitamin D (ergocalciferol 50,000 units every week)
  Other Names: Drisdol; Vitamin D
  Arms: Ergocalciferol
Drug: Placebo pill — The investigators will give control group 12 weeks of 1 placebo pill every week.
  Arms: Placebo pill

SUMMARY:
Recent clinical trials in non diabetics showed that vitamin D supplementation markedly reduced serum levels of C-reactive protein (CRP), interleukin-6, and tissue matrix metallo-proteinases. Our study objective is to evaluate if administration of vitamin D in African Americans with hypovitaminosis D and DM Type 2 decreases serum levels of inflammatory/thrombotic markers such as CRP: Highly Sensitive C Reactive Protein.

DETAILED DESCRIPTION:
Other questions in our study: In diabetic African American patients,

1. Prevalence of vitamin D deficiency?
2. Correlation/relationship between vitamin D levels, Calcium level, parathyroid hormone (PTH) and Inflammatory markers

Setting: All visits will take place at the Fantus Diabetes Clinic.

ELIGIBILITY:
Inclusion Criteria:

* African Americans
* DM type 2

Exclusion Criteria:

* symptomatic vitamin D deficiency
* hypocalcemia
* hypercalcemia
* malabsorption
* liver disease
* patients with creatinine > 1.5. (CKD >/= 3)
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-04; Primary Completion 2010-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Levels of inflammatory markers | baseline and 12 weeks

SECONDARY OUTCOMES:
Levels of Vitamin D, PTH and Calcium | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leon Fogelfeld, MD, Study Director — Cook County Health